CLINICAL TRIAL: NCT00044876
Title: Treatment of Leiomyomata With the Selective Progesterone Receptor Modulator CDB-2914
Brief Title: Treatment of Uterine Fibroids With CDB-2914, an Experimental Selective Progesterone Receptor Antagonist
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020287; 02-CH-0287
Record Dates: First submitted 2002-09-05; First posted 2002-09-06 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-10-01

CONDITIONS: Leiomyoma
Keywords: Endometrium; Progesterone; Estrogen; Leiomyoma; Uterine Leiomyoma; Uterine Fibroids; Fibroids
MeSH Terms: conditions — Leiomyoma; Myofibroma | interventions — ulipristal

INTERVENTIONS:
Drug: CDB-2914

SUMMARY:
Uterine leiomyomata (fibroids) are a common benign tumor of the uterine muscle in premenopausal women. These tumors may cause bleeding, pelvic pain and pressure. Because fibroids grow in the presence of estrogen, medical therapies that decrease estrogen levels (like GnRH analog) cause fibroids to shrink and so may relieve symptoms. However, such medication can only be given short-term and has inconvenient side effects such as hot-flushes. Thus, many women with symptomatic fibroids choose to have them removed surgically, either individually or by removing the uterus via hysterectomy.

The study evaluates a new medical treatment for fibroids using the progesterone receptor modulator CDB-2914. A similar compound, mifepristone (Registered Trademark), reduced fibroid size when given for twelve weeks. This study will compare fibroid size, hormone levels and symptoms before and during daily administration of CDB-2914 (10 or 25 mg) or placebo for 10 - 14 weeks. To do this, women will undergo MRI and a saline hysterosonogram (ultrasound with fluid) of the uterus before and at the end of the treatment; they will have blood drawn every 7 - 14 days, and will fill out a symptom calendar at home. Hysterectomy will be performed at the end of the treatment to evaluate the effects of the medication on the uterine and fibroid tissues, and to provide treatment for the study participant. Women will be randomly assigned to the treatment groups; during the treatment period neither the participants nor the investigators will know the type of treatment that a woman receives.

...

DETAILED DESCRIPTION:
Uterine leiomyomata (fibroids) are a common benign tumor of the uterine muscle in premenopausal women. These tumors may cause bleeding, pelvic pain and pressure. Because fibroids grow in the presence of estrogen, medical therapies that decrease estrogen levels (like GnRH analog) cause fibroids to shrink and so may relieve symptoms. However, such medication can only be given short-term and has inconvenient side effects such as hot-flushes. Thus, many women with symptomatic fibroids choose to have them removed surgically, either individually or by removing the uterus via hysterectomy.

The study evaluates a new medical treatment for fibroids using the progesterone receptor modulator CDB-2914. A similar compound, mifepristone (Registered Trademark), reduced fibroid size when given for twelve weeks. This study will compare fibroid size, hormone levels and symptoms before and during daily administration of CDB-2914 (10 or 25 mg) or placebo for 10 - 14 weeks. To do this, women will undergo MRI and a saline hysterosonogram (ultrasound with fluid) of the uterus before and at the end of the treatment; they will have blood drawn every 7 - 14 days, and will fill out a symptom calendar at home. Hysterectomy will be performed at the end of the treatment to evaluate the effects of the medication on the uterine and fibroid tissues, and to provide treatment for the study participant. Women will be randomly assigned to the treatment groups; during the treatment period neither the participants nor the investigators will know the type of treatment that a woman receives.

ELIGIBILITY:
* GENERAL INCLUSION CRITERIA:

Women receiving insulin or thyroid hormone replacement may participate if well-controlled; use of vitamins and calcium under RDA is allowed.

Female gender-to evaluate effects in the target population for clinical trials.

In good health. Chronic medication use is acceptable except for glucocorticoid use. Other chronic medication use may be acceptable at the discretion of the research team. Interval use of over-the counter drugs is acceptable but must be recorded.

Menstrual cycles of 24 - 35 days.

Hemoglobin greater than 10 g/dL.

Willing and able to comply with study requirements.

Age 33 to 50.

Using mechanical (condoms, diaphragms), sterilization or abstinence methods of contraception for the duration of the study.

Negative urine pregnancy test.

BMI less than or equal to 33.

Able to read and speak English fluently to allow accurate self-administration of medication, recording of symptoms and unassisted completion of questionnaire.

Normal glomerular filtration rate.

Liver function tests within 130% of upper limit.

INCLUSION CRITERIA FOR WOMEN WITH LEIOMYOMA:

History of uterine leiomyoma causing symptoms of bleeding, pressure, or pain, as defined by the ACOG practice bulletin (ACOG Practice Bulletin 1994):

Excessive uterine bleeding will be evidenced by either of the following-profuse bleeding with flooding or clots or repetitive periods lasting for more than 8 days; or anemia due to acute or chronic blood loss; OR

Pelvic discomfort caused by leiomyomata, either acute and severe or chronic lower abdominal or low back pressure or bladder pressure with urinary frequency not due to urinary tract infection.

Uterine leiomyoma(ta) of at least 2 cm size.

No desire for fertility; willing to undergo hysterectomy.

GENERAL EXCLUSION CRITERIA:

Significant abnormalities in the history, physical or laboratory examination.

Pregnancy.

Lactation.

Use of oral, injectable or inhaled glucocorticoids or megesterol within the last year.

Unexplained vaginal bleeding.

History of malignancy within the past 5 years.

Use of estrogen or progesterone-containing compounds, such as oral contraceptives and hormone replacement therapy, within 8 weeks of study entry, including transdermal, injectable, vaginal and oral preparations.

Use of agents known to induct hepatic P450 enzymes; use of imidazoles.

Current use of GnRH analogs or other compounds that affect menstrual cyclicity.

FSH greater than 20 IU/mL.

Significant medical disorders.

Cervical dysplasia.

Need for interval use of narcotics.

Abnormal adnexal/ovarian mass.

Intrauterine device.

EXCLUSION CRITERIA FOR WOMEN WITH FIBROIDS:

Use of herbal medication having estrogenic or antiestrogenic effects within the past 3 months.

Contradiction to anesthesia

Genetic causes of leiomyomata.

Previous participation in the study.

Known recent rapid growth of fibroids, defined as a doubling in size in six months.

Ages: 33 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2002-09-02; Primary Completion 2007-06-16 (Actual); Study Completion 2015-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynnette K Nieman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Batista MC, Cartledge TP, Zellmer AW, Merino MJ, Axiotis C, Loriaux DL, Nieman LK. Delayed endometrial maturation induced by daily administration of the antiprogestin RU 486: a potential new contraceptive strategy. Am J Obstet Gynecol. 1992 Jul;167(1):60-5. doi: 10.1016/s0002-9378(11)91627-5. PMID 1442957
- [Background] Cadepond F, Ulmann A, Baulieu EE. RU486 (mifepristone): mechanisms of action and clinical uses. Annu Rev Med. 1997;48:129-56. doi: 10.1146/annurev.med.48.1.129. PMID 9046951
- [Background] Burroughs KD, Howe SR, Okubo Y, Fuchs-Young R, LeRoith D, Walker CL. Dysregulation of IGF-I signaling in uterine leiomyoma. J Endocrinol. 2002 Jan;172(1):83-93. doi: 10.1677/joe.0.1720083. PMID 11786376
- [Derived] Wei Q, Levens ED, Stefansson L, Nieman LK. Indian Hedgehog and its targets in human endometrium: menstrual cycle expression and response to CDB-2914. J Clin Endocrinol Metab. 2010 Dec;95(12):5330-7. doi: 10.1210/jc.2010-0637. Epub 2010 Sep 29. PMID 20881264